CLINICAL TRIAL: NCT01320098
Title: Home-Based Parent Training in ADHD Preschoolers
Brief Title: Parent Training for Attention Deficit Hyperactivity Disorder (ADHD) Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01MH074556-04 (NIH)
Record Dates: First submitted 2011-03-11; First posted 2011-03-22 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention; Behavior Problems; Compliance; Evaluation; Preschool; ADHD; Overactive; Inattentive; Attention Deficit Hyperactivity Disorder in Preschoolers
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Home-Based Parenting Program (Experimental)
  Interventions: Behavioral: Home-Based Parenting Program
- Clinic-Based Parenting Program (Experimental)
  Interventions: Behavioral: Clinic-Based Parenting Program
- Wait-List Control Group (Other)
  Interventions: Behavioral: Wait-List Control Group

INTERVENTIONS:
Behavioral: Home-Based Parenting Program — The Home-Based Parenting Program aims to improve impulsive and oppositional behaviors in 3 and 4 year-olds. The program involves 8 home visits with a therapist. The visits focus on the skills listed below as a means of improving your child's behavior.
  1. Helping you set developmentally appropriate goals for your child. One way we do this is by focusing on situations that occur naturally in your home. Another way is by having you engage in activities with your child that focus on improving attention and the ability to delay.
  2. Increasing the quality and quantity of positive interactions between you and your child
  3. Changing the way you respond to your child's inappropriate behaviors so as to reduce the frequency of negative interactions.
  4. Improving your parenting skills. This program also includes between-session "homework tasks" so that you can practice the skills you have learned throughout the week.
  Arms: Home-Based Parenting Program
Behavioral: Clinic-Based Parenting Program — The Clinic-Based Parenting Program aims to improve ADHD symptoms by reducing noncompliance, which is common in children with ADHD. Parents learn how to help their child attend to and comply with requests and directions so as to improve compliance and attention.
  The program involves 8 clinic visits with a therapist. Parents learn various parenting skills to help improve their child's behaviors.
  Parents learn techniques and skills to promote positive interactions with their child, including:
  1. Increasing the positive attention you give to your child.
  2. Reducing the inappropriate use of commands, questions and criticisms.
  3. Appropriate use of praise and physical attention (e.g., hugs) as rewards.
  4. Actively ignoring minor, inappropriate behaviors. Parents also learn how to: increase compliance via clear instruction; respond to compliant and noncompliant behaviors; and create and use clear rules about appropriate and inappropriate child behaviors.
  Arms: Clinic-Based Parenting Program
Behavioral: Wait-List Control Group — If your child is randomized to the 8-week Wait-List group, you and your child will be asked to attend 2 assessment visits -1 screening/baseline visit and one 8 weeks later. These assessment visits will take place at our clinic. After completing the second assessment, you will receive your choice of either the home-based or clinic-based parenting program.
  Arms: Wait-List Control Group

SUMMARY:
The purpose of this research is to evaluate and compare the effectiveness of two parenting programs in reducing the ADHD symptoms and behavioral problems of preschool children with ADHD through a controlled study. One program is a home-based parent training intervention that is designed to enhance the parent-child interaction, constructive parenting skills, and the child's tolerance for delay. The other intervention is a clinic-based parent training program that focuses on reducing noncompliance in preschool children and improving parenting skills.

Both programs consist of private weekly parenting sessions with Clinical Psychologists - once a week for 8 weeks. The sessions are 1-1.5 hours in length. Both programs use behavior modification as a means of improving oppositional and non-compliant child behavior. Both interventions also involve procedures that focus on improving children's attention.

Neither program involves medication, and all families will receive one of the two parenting programs being evaluated. Study evaluations, as well as participation in the parenting programs, are provided at no cost to families. Evaluation and parenting sessions can be scheduled at times convenient to families.

ELIGIBILITY:
Inclusion Criteria:

* Age = 3.0 - 4.11
* In preschool program at least 2 half days per week
* Meets criteria for ADHD on clinical evaluation / DISC
* ADHD severity: > 1.5 SD above mean for age/sex on CTRS-R
* ADHD severity: > 1.0 SD above mean for age/sex on CPRS-R

Exclusion Criteria:

* Current Medication treatment for ADHD
* IQ < 70 (Full Scale on WPPSI III)
* Pervasive Developmental Disorder
* Psychosis
* Severe receptive language impairment
* Neurological Disorder
* Significant medical disorder
* Primary caretaker is not able to participate
* Non-English speaking primary care taker

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2007-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Conners Teacher Rating Scale | Post-Treatment (within one week of the last treatment session / end of the 8 week waiting period)
  Behavior Rating Scale

SECONDARY OUTCOMES:
Conners Parent Rating Scale | Post-Treatment (within one week of the last treatment session / end of the 8 week waiting period)
  Behavior Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Howard Abikoff, Ph.D., Principal Investigator — New York University Child Study Center
Locations (1):
- NYU Child Study Center, One Park Avenue, New York, New York, United States

REFERENCES:
- [Derived] Abikoff HB, Thompson M, Laver-Bradbury C, Long N, Forehand RL, Miller Brotman L, Klein RG, Reiss P, Huo L, Sonuga-Barke E. Parent training for preschool ADHD: a randomized controlled trial of specialized and generic programs. J Child Psychol Psychiatry. 2015 Jun;56(6):618-31. doi: 10.1111/jcpp.12346. Epub 2014 Oct 16. PMID 25318650
- See also: Related Info — http://www.aboutourkids.org/research/research_studies/recruiting_studies